CLINICAL TRIAL: NCT05532462
Title: Trans-nasal Complete Nasolabial Cyst Excision
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Ibrahim Yousef, Principal Investigator, Sohag University
Other Study IDs: SH_1180
Record Dates: First submitted 2022-08-24; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Nasolabial Cyst
Keywords: Nasoalveolar - Nasolabial - Klestadt's - Cyst

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Trans-nasal complete nasalabial cyst excision — The surgery is carried out mainly using x5 magnification loupe and 0° degree sinoscope. Submucosal infiltration (lidocaine 2% and 1:100,000 adrenaline). An incision was made at the mucosal covering of the cyst wall and nasal floor in a transverse and anteroposterior direction. The mucosal flap is elevated and separated from the cyst wall and reflected toward the septum side. During dissection, cyst content is usually drained. The whole cyst wall was carefully dissected with sharp and blunt dissection from the mucous membrane, and laterally from the premaxillary area. Finally, endoscopic examination to check the operative bed and refashioning mucosal flap coverage. If mucosal flap is lacerated, then excised and operative bed left for healing by creeping from surrounding edges. Endoscopic trans-nasal complete excision has a shorter operative time, minimal intraoperative bleeding, and no postoperative pain or edema reported.
  Other Names: sublabial approach

SUMMARY:
Background: Nasolabial cysts are rare benign epithelial nonodontogenic soft tissue cysts arising in the nasal alar region. Sublabial excision or transnasal endoscopic marsupialization is the standard treatment.

Patients and methods: Between 2019 and 2022, a descriptive retrospective study, including 20 patients who presented with Nasolabial cysts, was conducted.

DETAILED DESCRIPTION:
A retrospective study of patients who were presented in the period from 2019 to 2022, with nasolabial cysts. Patients' files were checked for demographic data, clinical presentation, preoperative radiological investigations, histopathology, surgical approach, complications, and outcome.

Technique:

The surgery is carried out mainly using x5 magnification loupe and 0° degree sinoscope. Submucosal infiltration (lidocaine 2% and 1:100,000 adrenaline). An incision was made at the mucosal covering of the cyst wall and nasal floor in a transverse and anteroposterior direction. The mucosal flap is elevated and separated from the cyst wall and reflected toward the septum side. During dissection, cyst content is usually drained. The whole cyst wall was carefully dissected with sharp and blunt dissection from the mucous membrane, and laterally from the premaxillary area. Finally, endoscopic examination to check the operative bed and refashioning mucosal flap coverage. If mucosal flap is lacerated, then excised and operative bed left for healing by creeping from surrounding edges. Endoscopic trans-nasal complete excision has a shorter operative time, minimal intraoperative bleeding, and no postoperative pain or edema reported.

ELIGIBILITY:
Inclusion Criteria:

•Nasolabial cyst

Exclusion Criteria:

* Recurrent cases
* Previous operated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In upper Egypt In sohag universiy hospital terriary center
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Symptoms and clinical sign | 2 years
  The presenting symptoms which made the patient sought medical advice
Preoperative Computer tomography or soft tissue ultrasound | 2 years
  Radiological description of the lesion
lining epithelium and inflammatory cell in wall of histopathology | 2 years
  histopathological criteria of the epithelium and cyst wall
complications and outcome | 2 years
  postoperative complication or recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed Elrabie Ahmed, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
A retrospective study of patients who were presented in the period from 2019 to 2022, with nasolabial cysts